CLINICAL TRIAL: NCT06906887
Title: PULSO Trial: Pulsed Low-Dose-Rate (PLDR) Radiation Chemoradiation (CRT) vs. Standard CRT for Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lindsay Puckett, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00049620
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer; Oesophageal Cancer; GastroEsophageal Cancer
Keywords: Pulsed Low-Dose-Rate Radiation; Chemoradiation; esophagitis; Esophagectomy; Esophageal Cancer; Oesophageal Cancer; GastroEsophageal Cancer; Pulsed reduced dose rate radiation; Pulsed radiation
MeSH Terms: conditions — Esophageal Neoplasms; Esophagitis | interventions — Induction Chemotherapy; Drug Therapy; Heart Rate; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pulsed Low-Dose-Rate Radiation (PLDR) (Experimental): Neoadjuvant radiation delivered in short pulses; same dose as standard chemoradiation arm.
  Interventions: Drug: Induction Chemotherapy (modified FLOT or modified FOLFOX-6); Drug: Chemotherapy; Radiation: Pulsed Low-Dose-Rate (PLDR) Radiation; Procedure: Surgery
- Standard Chemoradiation (Experimental): Standard (non-pulsed) neoadjuvant radiation; same dose as PLDR arm.
  Interventions: Drug: Induction Chemotherapy (modified FLOT or modified FOLFOX-6); Drug: Chemotherapy; Radiation: Conventional Radiation; Procedure: Surgery

INTERVENTIONS:
Drug: Induction Chemotherapy (modified FLOT or modified FOLFOX-6) — Subjects are expected to receive 2-4 months of induction chemotherapy; the interval and dosages will be determined and can be modified at the discretion of their medical oncologist. The preferred induction chemotherapies are modified FLOT or FOLFOX-6. Subjects can enroll if they receive less than 2 months of induction chemotherapy as long as they are deemed to be a candidate for concurrent chemoradiation therapy.
Drug: Chemotherapy — The preferred concurrent chemoradiation is carboplatin/paclitaxel weekly.
Radiation: Conventional Radiation — For both standard conventional radiation therapy and PLDR radiation therapy, the standard dose (5000cGy/25fx default, 4140-5040 in 23-28 fractions) should be given. Fractions should consist of 180-200 cGy per treatment.
  Arms: Standard Chemoradiation
Radiation: Pulsed Low-Dose-Rate (PLDR) Radiation — For both standard conventional radiation therapy and PLDR radiation therapy, the standard dose (5000cGy/25fx default, 4140-5040 in 23-28 fractions) should be given. Fractions should consist of 180-200 cGy per treatment.
  For PLDR radiation therapy, each fraction will be delivered as a series of 20 cGy (or 0.2 Gy) pulses that are separated by 3-minute time intervals.
  Arms: Pulsed Low-Dose-Rate Radiation (PLDR)
Procedure: Surgery — Esophagectomy is not required for trial and will be administered per medical judgement of the treating physicians. Surgery will take place at the time directed by the surgeon. This typically will take place approximately 6-13 weeks after chemoradiation therapy.

SUMMARY:
This is a prospective, randomized, open-label, two-arm phase 2 trial that will evaluate whether the use of Pulsed Low-Dose-Rate radiation technique, as compared to standard radiation, is associated with reduced rates of clinically significant esophagitis during and following chemoradiation.

DETAILED DESCRIPTION:
PLDR radiation technique has been shown to kill cancer cells while limiting normal tissue toxicity. In PLDR, subjects receive the same total dose of radiation for each treatment, but the treatment is delivered in a series of low-dose pulses which are separated by timed pauses. Radiation given with this approach may be less toxic but appears to be equally effective. This trial will evaluate the PLDR technique in combination with standard chemotherapy as part of definitive or curative treatment for locally advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

A potential study subject who meets all of the following inclusion criteria is eligible to participate in the study.

1. Age ≥ 18 years.
2. Stage II-IVb adenocarcinoma of the esophagus (if IVb, oligometastatic only, felt to be eligible for definitive dose CRT treatment by treating physician).
3. Currently receiving or have received induction chemotherapy and planned for definitive dose chemoradiation (+/- esophagectomy).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Adequate hematologic function within 30 days prior to registration defined as follows:

   1. Absolute Neutrophil Count ≥ 1,500/mcg
   2. Hemoglobin ≥ 8 gm/dL
   3. Platelets ≥ 100,000/mcL.
6. Adequate renal function within 30 days prior to registration, defined as a creatinine clearance of ≥ 50 ml/min as calculated by the Cockcroft-Gault equation.
7. Adequate hepatic function within 30 days prior to registration, defined as total bilirubin ≤ 1.5 x ULN

   a. Note: patients with known Gilbert Syndrome can have a total bilirubin < 2.5 x upper limit of normal (ULN).
8. Female patients <65 years of age and of childbearing potential must have a negative serum/urine pregnancy test within 14 days prior to study entry. A female not of childbearing potential is one who has undergone a hysterectomy, bilateral oophorectomy, tubal ligation, or who has had no menses for 12 consecutive months.
9. Patients of reproductive potential must agree to use effective contraception for the duration of study treatment. Effective contraception includes oral contraceptives, implantable hormonal contraception, double-barrier method, or intrauterine device.
10. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
11. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

A potential study subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Age < 18 years.
2. Extensive distant metastatic cancer, defined as >5 metastases.
3. Recurrent esophageal cancer.

   a. Note: prior or concurrent malignancies are allowed if they do not impact the study's primary endpoint (i.e., treatment-associated toxicity).
4. Prior non-approved chemotherapy for the treatment of cancer.
5. Prior radiotherapy to the region of the study cancer that would result in an overlap of radiation therapy fields.
6. Women must not be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
New prescription for narcotics | Up to 6 weeks after radiation treatment
  The number of subjects requiring a new prescription for narcotics.
Increasing existing narcotics | Up to 6 weeks after radiation treatment
  The number of subjects increasing existing narcotics by 25%.
Oral intake | Up to 6 weeks after radiation therapy
  The number of subjects transitioning from solid to liquid or liquid to no oral intake.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Puckett, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No